CLINICAL TRIAL: NCT02544009
Title: Quantifying Weight Regain and the Persistence of Metabolic Adaptation Following Extreme Weight Loss
Brief Title: Quantifying the Persistence of Metabolic Adaptation and Weight Regain Following Extreme Weight Loss
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150192; 15-DK-0192
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Energy Expenditure
Keywords: Energy Expenditure; Obesity; Behavioral Weight Loss Treatment; Natural History
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: 16 subjects who previously participated in the Biggest Loser study

SUMMARY:
Background:

Many people regain the weight they lose through diet and exercise. This might happen because the weight loss slows their metabolism. This slowing is called metabolic adaptation. It may cause people to regain weight if they do not keep up high levels of exercise or major caloric restrictions. Researchers want to find the long-term effects of metabolic adaptation in the previous Biggest Loser study participants. They hope to learn the body s response to lifestyle changes that result in weight loss. They also want to see if certain changes can lead to longer-term success in maintaining weight loss.

Objectives:

To better understand the long-term metabolic changes caused by rapid weight loss achieved through diet restriction and vigorous physical activity.

Eligibility:

Former Biggest Loser research study participants (Protocol No. PBRC29008).

Design:

Participants will be screened with a phone interview.

This study has 3 phases.

Phase 1 will last at least 3 weeks. Participants will receive a physical activity monitor and wireless scale. These will send their daily weight and activity back to NIH.

In Phase 2, participants will stay at NIH for 3 days. Their metabolism will be measured through:

Their activity monitor

Urine samples and daily body weight

Medical review and physical exam

Fasting for 12 hours each night for a blood draw the following morning

DEXA: a low-dose x-ray of the body

BIS: Electrodes on the hand/wrist and foot/ankle measure body water content.

Phase 3 will last at least 3 weeks. Participants will:

Continue to monitor their daily weight and activity

Collect urine samples and send them back to NIH

DETAILED DESCRIPTION:
Weight loss is accompanied by a slowing of metabolic rate. Metabolic slowing often occurs to a degree greater than predicted by the amount of weight lost, a phenomenon called metabolic adaptation , and is hypothesized to persist over time and promote weight regain. We previously discovered large metabolic adaptations in response to the intensive lifestyle intervention as part of The Biggest Loser weight loss competition. Those subjects rapidly lost massive amounts of weight and their resting energy expenditure decreased by ~500 kcal/d more than was expected based on their body composition at the end of the intervention. The purpose of this study is to investigate whether the metabolic adaptation has persisted in the years following the intervention in the same subjects. Furthermore, we will measure body weight and composition in these subjects and investigate the correlates of weight regain.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 16 subjects who previously participated in the Biggest Loser study (Pennington Biomedical Research Center protocol no. PBRC29008).
* Written informed consent

EXCLUSION CRITERIA:

* Volunteers unwilling or unable to give informed consent.
* Women who are pregnant or breastfeeding cannot participate in the study. A pregnancy test will be performed during the first day of the inpatient visit. If the pregnancy test is positive, the subject cannot continue to participate in the study.
* Subjects with implantable cardio-defibrillator or pacemaker may not participate in the bioelectric impedance spectroscopy (BIS) testing portion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This natural history study includes enrollment of 16 adult subjects who previously participated in the Biggest Loser intervention and participated in a study of body composition and metabolic changes [1]. Several years following weight loss intervention, these subjects may have experienced weight regain and either persistence or remission of the previously observed metabolic adaptation. The present study was designed to investigate the persistence of metabolic adaptation and explore whether the degree of metabolic adaptation during the weight loss intervention was correlated with body weight and body fat regain.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-09-05; Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Measure body composition and REE several years after completion of The Biggest Loser intervention. Metabolic adaptation will be calculated as the difference between the measured REE and the REE predicted from linear regression analysis of baseli... | 2 weeks
  The primary analysis will use a t-test to test the null hypothesis that this difference is equal to zero. Secondary analyses will explore predictors of metabolic adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Kerns JC, Guo J, Fothergill E, Howard L, Knuth ND, Brychta R, Chen KY, Skarulis MC, Walter PJ, Hall KD. Increased Physical Activity Associated with Less Weight Regain Six Years After "The Biggest Loser" Competition. Obesity (Silver Spring). 2017 Nov;25(11):1838-1843. doi: 10.1002/oby.21986. PMID 29086499
- [Derived] Fothergill E, Guo J, Howard L, Kerns JC, Knuth ND, Brychta R, Chen KY, Skarulis MC, Walter M, Walter PJ, Hall KD. Persistent metabolic adaptation 6 years after "The Biggest Loser" competition. Obesity (Silver Spring). 2016 Aug;24(8):1612-9. doi: 10.1002/oby.21538. Epub 2016 May 2. PMID 27136388
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0192.html